CLINICAL TRIAL: NCT03207113
Title: Adoption, Acceptability, and Effectiveness of a Mobile Health App for Personalised Prostate Cancer Survivorship Care: a Realist Case Study of the Ned App.
Brief Title: Adoption, Acceptability, and Effectiveness of a Mobile Health App for Personalised Prostate Cancer Survivorship Care.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Global eHealth Innovation (Other)
Collaborators: Trillium Health Partners (Other); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: THP REB ID#826
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
Keywords: prostate-specific antigen; prostate cancer survivorship; mobile health; realist evaluation; case study
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ned Group (Experimental): Participants in the Ned case study (patients, caregivers, clinicians) will receive access to the Ned application.
  Ned ("No Evident Disease") is the first application to provide patients with access to individual-level prostate-specific antigen values streamed directly from the Ontario Laboratory Information System to their own smartphone. The application aims to promote self-care by informing patients directly of their PSA results and providing them with a personalised view of their own symptoms. It supports real-time clinical decision-making by providing clinicians with patient-reported outcomes collected in-app, and includes a curated educational feed and support group links.
  Interventions: Behavioral: Ned

INTERVENTIONS:
Behavioral: Ned — Prostate cancer survivorship application.

SUMMARY:
The Ned case study is a 12-month mixed methods embedded single-case study with a nested within-group pre-post comparison of health outcomes. 400 patients, 200 caregivers, and 10 clinicians will be given access to Ned. Participants will be asked to complete study assessments at baseline, 2 months, 6 months and 12 months. 30 semi-structured qualitative interviews with patients (n=20) and their caregivers (n=10) post-study will also be conducted to gain insight into their experience with the application.

DETAILED DESCRIPTION:
By 2030, prostate cancer will be the most commonly diagnosed cancer in North America. To mitigate this impending challenge, comprehensive support mechanisms for disease and treatment-specific changes in health and wellbeing must be proactively designed and thoughtfully implemented for streamlined survivorship care. Mobile health applications have been lauded as a promising complement to current outpatient treatment and monitoring strategies, but have not yet been widely used to support prostate cancer survivorship needs. A realist evaluation is needed to examine the impact of such applications on the prostate cancer survivorship experience.

The investigators seek to gain an understanding of how a mobile health application for prostate cancer survivorship care called Ned ("No Evident Disease") is adopted and accepted by patients, caregivers and clinicians. The investigators also aim to determine the effect of Ned on health-related quality of life, satisfaction with cancer care, unmet needs, self-efficacy, and prostate cancer-related levels of anxiety.

The Ned case study is a 12-month mixed methods embedded single-case study with a nested within-group pre-post comparison of health outcomes. 400 patients, 200 caregivers, and 10 clinicians will be given access to Ned. Participants will be asked to complete study assessments at baseline, 2 months, 6 months and 12 months. 30 semi-structured qualitative interviews will be conducted with patients (n=20) and their caregivers (n=10) post-study to gain insight into their experience with the application.

This will be the first realist case study to evaluate an application for prostate cancer survivorship care. Prostate cancer survivors are set to increase in number and longevity, heightening the need for integrated survivorship solutions to provide them with optimal and durable outcomes. The knowledge gained from this study will comprehensively inform how and why Ned works, for whom, and in what circumstances. Understanding the impact of digital health interventions like Ned on how survivors care for themselves is critical to realising patient-centered care.

ELIGIBILITY:
Patients must meet the following eligibility criteria to be enrolled into the study:

* 18 years of age or older
* Receiving care at the THP Mississauga Hospital or Credit Valley Hospital
* Pathology report confirming prostate cancer diagnosis via transrectal, transperineal or transurethral biopsy (standard 12-core template)
* Life expectancy > 1 year
* No concomitant cancer diagnosis
* Own a device that is compatible with the Ned application and is web-enabled through a data plan and/or wifi capabilities (e.g. laptop, desktop, tablet, smartphone)
* Able to read, write and speak English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Adoption | Continuous throughout 12 month study duration
  The number of patients, caregivers and clinicians who are invited to open a Ned account, and the consequent number of Ned accounts created; measured using analytics log data.
Acceptability | Continuous throughout 12 month study duration
  The perception of Ned as an acceptable addition to the standard of care; measured using (i) analytics log data (ii) validated questionnaires (iii) semi-structured interviews.

SECONDARY OUTCOMES:
Health-related quality of life | 12 month study duration
  Health-related quality of life will be measured using a validated questionnaire. Data will be collected at baseline, 2 months, 6 months, and 12 months.
Satisfaction with cancer care | 12 month study duration
  Satisfaction with cancer care will be measured using a validated questionnaire. Data will be collected at baseline, 2 months, 6 months, and 12 months.
Unmet needs | 12 month study duration
  Unmet needs will be measured using a validated questionnaire. Data will be collected at baseline, 2 months, 6 months, and 12 months.
Self-efficacy | 12 month study duration
  Self-efficacy will be measured using a validated questionnaire. Data will be collected at baseline, 2 months, 6 months, and 12 months.
Prostate cancer-related levels of anxiety | 12 month study duration
  Prostate cancer-related levels of anxiety will be measured using a validated questionnaire. Data will be collected at baseline, 2 months, 6 months, and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Feifer, MD, MPH, Principal Investigator — Trillium Health Partners
Locations (1):
- Centre for Global eHealth Innovation, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ned website. — http://getned.com